CLINICAL TRIAL: NCT02276820
Title: A Phase I Study Using Most Closely HLA-matched Adenovirus-specific T Lymphocytes for the Treatment of Adenovirus Infections Post-allogeneic Stem Cell Transplant(VIRALYM-A)
Brief Title: Most Closely Human Leukocyte Antigen (HLA)-Matched Adenovirus-specific T Lymphocytes (Viralym-A)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor is pursuing a different product for this indication
Sponsor: AlloVir (Industry)
Collaborators: Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H35136 Viralym-A; 5406 (Other: OPD)
Record Dates: First submitted 2014-10-20; First posted 2014-10-28 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Adenovirus Infection
Keywords: Adenovirus; Virus specific T cells; Viral infections
MeSH Terms: conditions — Adenoviridae Infections; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Viralym-A (Experimental): Partially HLA-matched Viralym-A cells will be thawed and given by intravenous injection. Patients will receive 2 x 10^7 partially HLA-matched Viralym-A/m2 as a single infusion.
  If a patient has a partial response they are eligible to receive up to 4 additional doses at biweekly intervals. These doses would come from the original infused line if sufficient vials were available but may come from another line if there are insufficient cells in the original line.
  Interventions: Biological: Viralym-A

INTERVENTIONS:
Biological: Viralym-A — Follow-up Assessments: The timing of follow-up visits is based on the date of Viralym-A infusion. If a patient has multiple Viralym-A infusions the schedule resets again at the beginning so follow up relates to the last Viralym-A infusion.
  Follow up will occur at 7 days, 14 days, 21 days, 28 days, 42 days, 90 days, 180 days, and 365 days post enrollment.
  Other Names: AdV-specific T cells

SUMMARY:
Patients enrolled on this study will have received a stem cell transplant. After a transplant, while the immune system grows back the patient is at risk for infection. Some viruses can stay in the body for life, and if the immune system is weakened (like after a transplant), they can cause life-threatening infections.

Adenovirus (AdV) is a virus that just causes symptoms of a common cold normally, but which can cause serious life-threatening infections in patients who have weak immune systems. It usually affects the lungs and can cause a very serious pneumonia, but it can also affect the gut, the liver, the pancreas and the eyes.

Investigators want to see if they can use a kind of white blood cell called T cells to treat adenovirus infections that occur after a transplant. Investigators have observed in other studies that treatment with specially trained T cells has been successful when the cells are made from the transplant donor. However as it takes 1-2 months to make the cells, that approach is not practical when a patient already has an infection.

Investigators have now generated AdV-specific T cells from the blood of healthy donors and created a bank of these cells. Investigators have previously successfully used frozen virus-specific T cell lines generated from healthy donors to treat virus infections after bone marrow transplant, and have now improved the production method and customized the bank of lines to specifically and exclusively target AdV.

In this study, investigators want to find out if the banked AdV-specific T cells derived from healthy donors are safe and can help to treat adenoviral infection.

The AdV-specific T cells (Viralym-A) are an investigational product not approved by the Food and Drug Administration (FDA).

Funding source - FDA OOPD

DETAILED DESCRIPTION:
To make AdV-specific T cells (Viralym-A cells), small pieces of protein called peptides that come from AdV were mixed with blood cells from healthy donors. These peptides train a kind of white blood cell called T cells to recognize and kill cells that are infected with AdV. These T cells were then grown in special growth factors in special flasks in the lab. Once we made sufficient numbers of cells, we tested them to make sure they recognized cells infected by adenovirus, and then we froze them.

When we think the subject needs them, Viralym-A cells will be thawed and injected into the intravenous line. To prevent an allergic reaction, prior to receiving Viralym-A cells the subject may be given diphenhydramine (Benadryl) and acetaminophen (Tylenol). The subject will remain in the clinic for at least one hour after the infusion. After the subject receives the cells, the transplant doctor will monitor the levels of adenovirus in the blood. We will also take blood to see how long the cells we gave the subject are lasting in the body.

Subjects will continue to be followed by their transplant doctors after the injection. The subject will either be seen in the clinic or they will be contacted by a research nurse to follow up for this study every week for 6 weeks, then at 3, 6 and 12 months. The subject may have other visits for their standard care. Subjects will also have regular blood tests done to follow their counts and the viral infection as part of their standard care.

To learn more about the way Viralym-A cells are working in the body, an extra 30-40 ml (6-8 teaspoons) of blood will be taken before the infusion and then at study follow-up visits at 1, 2, 3, 4 and 6 weeks, and 3 months after the infusion. Blood should come from the central intravenous line, and should not require extra needle sticks.

All participants on this study will be infused with the same number (dose) of cells. If Viralym-A infusion has helped the subjects infection or if they have had a treatment, for example with steroid drugs that might have destroyed the T cells the subject was given, then they are allowed to receive up to 4 additional infusions of the Viralym-A cells at the same initial dose level from 28 days after their initial infusion. Following infusions should be at least 14 days apart. After each Viralym-A cells infusion, subjects will be monitored as described above.

ELIGIBILITY:
Inclusion Criteria:

1. Prior myeloablative or non-myeloablative allogeneic hematopoietic stem cell transplant using either bone marrow or peripheral blood stem cells or single or double cord blood within 24 months.
2. Persistent or recurrent adenovirus infection or disease despite at least 7 days of standard therapy or failure of therapy as described below or if unable to tolerate standard therapy. Standard therapy is defined as antiviral therapy with cidofovir or an alternative antiviral agent if patient will not tolerate cidofovir therapy because of poor renal function.

   i. Adenovirus infection: defined as the presence of adenoviral positivity as detected by polymerase chain reaction (PCR) or culture from ONE site, such as stool or blood or urine or nasopharynx.

   ii. Adenovirus disease: defined as the presence of adenoviral positivity as detected by PCR, Direct fluorescent assay (DFA) or culture from two or more sites such as stool or blood or urine or nasopharynx.

   iii. Failure of therapy: defined as a rise or a fall of less than 50% in viral load in peripheral blood or any site of disease as measured by PCR (or any other quantitative assay) after 7 days of antiviral therapy.
3. Patients with multiple viral infections including AdV are eligible if their AdV infection is persistent despite standard therapy as defined above. Patients with multiple infections with one or more reactivation and one or more controlled infection are eligible to enroll.
4. Clinical status at enrollment to allow tapering of steroids to equal or less than 0.5 mg/kg/day prednisone (or equivalent).
5. Received transplant care locally and will remain in the Houston area for at least 6 weeks post Viralym-A infusion.
6. Hemoglobin (Hgb) > 8.0 (may be transfused).
7. Available Viralym-A T cell line.
8. Negative pregnancy test in female patients if applicable (childbearing potential who have received a reduced intensity conditioning regimen).
9. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

Exclusion Criteria:

1. Patients receiving Anti-thymocyte globulin (ATG), Campath or other immunosuppressive T cell monoclonal antibodies within 28 days of treatment with Viralym-A.
2. Patients with other uncontrolled/progressing infections defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to enrollment. For fungal infections patients must be receiving definitive systemic anti-fungal therapy and have no signs of progressing infection for 1 week prior to enrollment. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
3. Patients who have received donor lymphocyte infusion (DLI) within 28 days of Viralym-A infusion.
4. Requirement for FiO2 > 0.5 to maintain arterial oxygen saturation > 90%
5. Endotracheal intubation and mechanical ventilation at any FiO2
6. Hemodynamic instability requiring continuous infusions of inotropes or vasopressors
7. Patients who have received other investigational drugs within 28 days of Viralym-A infusion.
8. Patients with active acute graft versus host disease (GVHD) grades II-IV.
9. Active and uncontrolled relapse of malignancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of patients with adverse events after Viralym-A infusion | 42 days
  To determine if administration of banked AdV-specific T cells (Viralym-A) derived from healthy donors are safe in patients with AdV infection after allogeneic stem cell transplant.

SECONDARY OUTCOMES:
Assessment of adenoviral load response to the Viralym-A infusion | 1 year
  Viral load over time within a patient will be visualized to reveal the temporal patterns of immune response. Plots of smooth curves will be generated for each patient to graphically illustrate the pattern and duration of T-cell changes.
Reconstitution of antiviral immunity after Viralym-A infusion | 3 months
  Reconstitution of antiviral immunity over time within a patient will be visualized to reveal the temporal patterns of immune response. Plots of smooth curves will be generated for each patient to graphically illustrate the pattern and duration of T-cell changes.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Ramos, MD, Principal Investigator — Baylor College of Medicine; Swati Naik, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Childrens Hospital, Houston, Texas
  - The Methodist Hospital system, Houston, Texas

REFERENCES:
- [Background] Leen AM, Bollard CM, Mendizabal AM, Shpall EJ, Szabolcs P, Antin JH, Kapoor N, Pai SY, Rowley SD, Kebriaei P, Dey BR, Grilley BJ, Gee AP, Brenner MK, Rooney CM, Heslop HE. Multicenter study of banked third-party virus-specific T cells to treat severe viral infections after hematopoietic stem cell transplantation. Blood. 2013 Jun 27;121(26):5113-23. doi: 10.1182/blood-2013-02-486324. Epub 2013 Apr 22. PMID 23610374
- [Background] Papadopoulou A, Gerdemann U, Katari UL, Tzannou I, Liu H, Martinez C, Leung K, Carrum G, Gee AP, Vera JF, Krance RA, Brenner MK, Rooney CM, Heslop HE, Leen AM. Activity of broad-spectrum T cells as treatment for AdV, EBV, CMV, BKV, and HHV6 infections after HSCT. Sci Transl Med. 2014 Jun 25;6(242):242ra83. doi: 10.1126/scitranslmed.3008825. PMID 24964991